CLINICAL TRIAL: NCT05429736
Title: SCIMS Site Specific Project: Activating Spinal Circuits to Improve Walking, Balance, Strength, and Reduce Spasticity
Brief Title: Activating Spinal Circuits to Improve Walking, Balance, Strength, and Reduce Spasticity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edelle Field-Fote, PT, PhD, Principal Investigator, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1842303
Record Dates: First submitted 2022-05-02; First posted 2022-06-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Incomplete Spinal Cord Injury; Spasticity, Muscle
Keywords: spinal; cord; incomplete; motor; skill; training; transcutaneous; stimulation; TSS; tSCS; electrophysiology
MeSH Terms: conditions — Muscle Spasticity; Cone-Rod Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MST + TSS (Experimental): Individuals will participate in 6 training sessions of MST combined with TSS.
  Interventions: Behavioral: Motor Skill Training (MST); Device: Transcutaneous Spinal Stimulation (TSS)
- MST + ShamTSS (Sham Comparator): Individuals will participate in 6 training sessions of MST while receiving shamTSS.
  Interventions: Behavioral: Motor Skill Training (MST)

INTERVENTIONS:
Behavioral: Motor Skill Training (MST) — During MST participants will perform a series of 6 motor skill exercises designed to challenge balance, lower extremity coordination, agility, and speed. Five of these activities will be performed while standing to promote upright control and one activity will be performed while seated (alternating toe-tapping) to provide opportunity for active recovery. Participants will perform each exercise for one minute each, until 4 cycles of the circuit have been completed (approximately 45 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). During MST, participants will wear a chest-worn heart rate monitor to ensure that the optimal HRR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
Device: Transcutaneous Spinal Stimulation (TSS) — TSS will be delivered using a commercially available neuromuscular electrical stimulator. The active electrode will be positioned directly over the spine at the T11/T12 spinous interspace, and the reference electrode will be positioned over the umbilicus. Stimulation intensity will be gradually increased until paresthesia of the lower legs and feet is achieved or to the highest level each participant can tolerate. Stimulation will be delivered for a total duration of 30 min after paresthesia/ maximum tolerability is reached.
  Other Names: tSCS
  Arms: MST + TSS

SUMMARY:
For many people with spinal cord injury (SCI), the goal of walking is a high priority. There are many approaches available to restore walking function after SCI; however, these approaches often involve extensive rehabilitation training and access to facilities, qualified staff, and advanced technology that make practicing walking at home difficult. For this reason, developing training approaches that could be easily performed in the home would be of great value. In addition, non-invasive spinal stimulation has the potential to increase the effectiveness of communication between the brain and spinal cord. Combining motor skill training (MST) with transcutaneous spinal stimulation (TSS) may further enhance the restoration of function in persons with SCI. Therefore, the purpose of this study is to determine if moderate-intensity, MST can improve walking-related outcomes among persons with SCI and to determine if the addition of non-invasive TSS will result in greater improvements in function compared to training alone.

DETAILED DESCRIPTION:
Individuals with SCI will be asked to participate in this study over a four-week period. During the first 2 weeks (wash-in phase), individuals will participate in 6 aerobic and exercise training sessions as part of either an existing outpatient clinical program or by completing a personalized exercise plan. During the intervention phase (last 2 weeks), participants will be randomized to complete 6 training sessions of: 1) motor skill training combined with TSS (MST+TSS group) or 2) motor skill training combined with shamTSS (MST+shamTSS). All participants will complete 3 testing sessions: baseline testing 1 (prior the wash-in phase), testing 2 (after the completion of the wash-in phase and prior the intervention phase), and testing 3 (after the completion of the intervention phase) to assess their walking ability, balance, strength, and spasticity. During the intervention phase and to monitor within-session changes, participants will also complete a short version of walking function and balance assessments prior to and after each training session.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-70 years of age
* Have a spinal cord injury (neurological level C3-T12) that occurred ≥3 months (sub-acute to chronic) prior to enrollment
* Have ISNCSCI severity classification C or D
* Able to stand for at least 5 minutes (with or without the aid of an assistive device)
* Able to move each leg independently for at least 3 steps (with or without the aid of an assistive device)
* Able to rise from sit to stand with moderate assistance from one person
* Use of prescription medication(s) for control of spasticity if the dosage has not changed in the last 2 weeks and you notify the study staff if your medication(s) change during study participation
* Ability and willingness to consent and authorize use of personal health information
* Ability to follow multiple instructions and communicate pain or discomfort

Exclusion Criteria:

* Progressive spinal lesions including degenerative, or progressive vascular disorders of the spine and/or spinal cord
* Injuries below the neurological spinal level of T12
* Pregnant, or if you have reason to believe you are or may become pregnant due to unknown risks to the fetus associated with TSS
* History of cardiovascular irregularities
* Presence of orthopedic conditions that would adversely affect participation in exercise
* Implanted stimulators of any type will be excluded due to unknown potential of electrical stimulation effects (e.g., baclofen pump, epidural spinal stimulator, implanted cardiac defibrillator, diaphragmatic pacemaker)
* Any cuts or sensitivity of the skin near the level of stimulation
* Active cancer or history of cancer
* Inability and unwillingness to consent and authorize use of personal health information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in 10 Meter Walk Test | Testing 1(Day 1), Testing 2 (Day 12), Pre/Post Training 1-6 (Days 15, 17, 19, 22, 24, 26), Testing 3 (Day 27)
  Walking speed (as determined by the 10MWT) is the primary outcome measure for assessing walking function. Participants will complete 3 10MWT trials at each testing session, separated by 2 minutes of seated rest. The average walking speed of the 3 walks will be calculated and used in the analyses.

SECONDARY OUTCOMES:
Change of Spatiotemporal Gait Characteristic (Cadence) | Testing 1(Day 1), Testing 2 (Day 12), Pre/Post Training 1-6 (Days 15, 17, 19, 22, 24, 26), Testing 3 (Day 27)
  Gait quality will be assessed from spatiotemporal gait characteristics (cadence [strides/min], stride length [cm] of the weaker and stronger limbs, and step length symmetry) collected via instrumented walkway as participants completed three, 10MWT trials at each testing session. The average cadence across three walks will be used in the analysis.
Change of Spatiotemporal Gait Characteristic (Stride Length - Both Lower Extremities) | Testing 1(Day 1), Testing 2 (Day 12), Pre/Post Training 1-6 (Days 15, 17, 19, 22, 24, 26), Testing 3 (Day 27)
  Gait quality will be assessed from spatiotemporal gait characteristics (cadence [strides/min], stride length [cm] of the weaker and stronger limbs, and step length symmetry) collected via instrumented walkway as participants completed three, 10MWT trials at each testing session. The average stride length across three walks will be used in the analysis.
Change of Spatiotemporal Gait Characteristic (Step Length Symmetry - Symmetry Index) | Testing 1(Day 1), Testing 2 (Day 12), Training 1-6 (Days 15, 17, 19, 22, 24, 26), Testing 3 (Day 27)
  Gait quality will be assessed from spatiotemporal gait characteristics (cadence [strides/min], stride length [cm] of the weaker and stronger limbs, and step length symmetry) collected via instrumented walkway as participants completed three, 10MWT trials at each testing session. The average step length for each leg across three walks will be used to compute the symmetry index (%).
Change of Berg Balance Scale | Testing 1 (Day 1), Testing 2 (Day 12), Pre/Post Training 1-6 (Days 15, 17, 19, 22, 24, 26), Testing 3 (Day 27)
  Balance will be measured using the BBS. The BBS total score will be calculated for each participant at each testing session. The total range of scores for the BBS equals 0-56, with higher scores from baseline indicating greater balance performance and lower scores from baseline indicating worsened balance performance. A subset of the BBS will be assess before and after each training session.
Change of Falls Efficacy Scale-International Version (FES-I) | Testing 1 (Day 1), Testing 2 (Day 12), Testing 3 (Day 27)
  The FES-I total score will be calculated for each participant at each testing session to measure fear of falling. The total range of scores for the FES-I equals 16-64, with lower scores indicating decreased fear of falling.
Change of Spinal Cord Assessment Tool for Spastic Reflexes | Testing 1 (Day 1), Testing 2 (Day 12), Testing 3 (Day 27)
  The SCATS will be used to assess spasticity. The total range of scores possible for the SCATS is 0-18, with a total score of 0 indicating no lower limb spasticity and higher total scores indicating greater spasticity severity.
Change of Modified 5-Times Sit-to-Stand | Testing 1 (Day 1), Testing 2 (Day 12), Testing 3 (Day 27)
  The modified 5-times sit-to-stand test will be used as a measure of functional lower extremity strength. The average time to complete the test will be calculated at each testing session.
Change of 2 Minute Walk Test | Testing 1(Day 1), Testing 2 (Day 12), Testing 3 (Day 27)
  Functional walking capacity will be measured based on the 2MWT distance. Total distance walked in 2-minutes will be recorded for each participant at each testing session.
Change of Maximal Isometric Strength | Testing 1(Day 1), Testing 2 (Day 12), Testing 3 (Day 27)
  Knee extensor (quadriceps) and ankle plantar flexors (gastrocnemius and soleus) strength will be measured using an isokinetic dynamometer. Maximum knee extensor force will be analyzed based on the maximum force produced over three attempts.
Change of Torque vs Speed Production | Testing 1(Day 1), Testing 2 (Day 12), Testing 3 (Day 27)
  Torque vs speed production will be using an isokinetic dynamometer. Maximum rate of torque production will be calculated based on the highest rate measured over three attempts.
Change of Modified Spinal Cord Injury Spasticity Evaluation Tool (modified SCI-SET) | Testing 1 (Day 1), Testing 2 (Day 12), Testing 3 (Day 27)
  The modified SCI-SET is a subjective measure used to assess the effects of spasticity on daily life in people with SCI. It requires participants to recall their past 7 days when rating the impact of spasticity. The scale uses a range of -2 (very problematic) to +1 (helpful).

CONTACTS AND LOCATIONS:
Overall Officials: Edelle Field-Fote, PT, PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No